CLINICAL TRIAL: NCT04066764
Title: An Efficacy and Safety Study of New Oral Anticoagulants and Vitamin K Antagonists for the Anticoagulation for the Implantation of Vena Cava Filters: A Prospective Randomized Controlled Trial
Brief Title: Rivaroxaban and Vitamin K Antagonists for the Anticoagulation for the Implantation of Vena Cava Filters
Acronym: EPICT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Sir Run Run Shaw Hospital (Other); Huadong Hospital (Other); Shanghai Zhongshan Hospital (Other); Shanghai 5th People's Hospital (Other); Yantai Yuhuangding Hospital (Other); Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Zhenjie Liu, Principal Investigator, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHZhejiangU-002
Record Dates: First submitted 2019-08-22; First posted 2019-08-26 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Venous Thromboembolism
Keywords: venous thromboembolism; rivaroxaban; vena cava filters
MeSH Terms: conditions — Venous Thromboembolism | interventions — Rivaroxaban; Warfarin; Nadroparin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban (Experimental): Participants will receive rivaroxaban 15mg oral twice daily for 3 weeks after operation, later rivaroxaban 20mg oral once daily until 3 months after the filter is retrieved.
  Interventions: Drug: Rivaroxaban
- Warfarin/ Nadroparin (Active Comparator): Participants will receive Nadroparin 1mg/kg twice daily (subcutaneous), plus warfarin 3mg oral once daily for 5 days after the operation, later warfarin(oral) at individually titrated doses(0.75mg to 18mg) to achieve a target international normalized ratio (INR) of 2.0 to 3.0, once daily until 3 months after the filter is retrieved.
  Interventions: Drug: Warfarin; Drug: Nadroparin

INTERVENTIONS:
Drug: Rivaroxaban — 15mg twice daily for 3 weeks after operation, later 20mg once daily until 3 months after the filter is removed. Application: oral
  Other Names: Xarelto
  Arms: Rivaroxaban
Drug: Warfarin — 3mg for 5 days after the operation, later 0.75mg to 18mg depending on INR (2.0-3.0) until until 3 months after the filter is removed. Frequency: once daily Application: oral
  Other Names: coumadin
  Arms: Warfarin/ Nadroparin
Drug: Nadroparin — Dose: 1mg/kg Duration: 5 days after the operation Frequency: twice daily Application: subcutaneous
  Other Names: Fraxiparin
  Arms: Warfarin/ Nadroparin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of new oral anticoagulants and vitamin K antagonists for the anticoagulation for the implantation of vena cava filters in patients with deep venous thrombosis.

DETAILED DESCRIPTION:
Deep vein thrombosis (DVT) of lower extremities is a venous reflux disorder caused by abnormal coagulation of deep vein blood. The main adverse consequences of DVT are pulmonary embolism (PE) and post-thrombotic syndrome, which can significantly affect the quality of life of patients and even lead to death. Anticoagulation is the basic treatment of DVT, which can inhibit the spread of thrombus, facilitate thrombus autolysis and recanalization of the lumen, and reduce the incidence and mortality of PE. For patients with contraindications or complications of anticoagulation therapy, the implantation of inferior vena cava filter may be considered. At the same time, patients with the following conditions may be considered for the implantation of inferior vena cava filter: PE is still present in the case of adequate anticoagulant therapy, floating thrombus in the iliac, femoral or inferior vena cava, thrombectomy is planned for acute DVT, and abdominal, pelvic or lower extremity surgery with high risk factors for PE and acute DVT. The current standard treatment regimen for venous thromboembolism (VTE) anticoagulation is low molecular weight heparin (LMWH) combined with or followed by vitamin K antagonist warfarin. It has been proved that low molecular weight heparin has good safety and effectiveness in the prevention and initial treatment of VTE, especially for VTE prevention and treatment in cancer patients and pregnant patients. As a standard oral anticoagulant, warfarin has definite anticoagulant effect and is cheap. However, low molecular weight heparin needs subcutaneous injection, which can cause adverse reactions such as pain, itching, subcutaneous hemorrhage and nodules at the injection site, and some complications such as heparin-induced thrombocytopenia (HIT). Warfarin anticoagulation therapy requires long-term laboratory monitoring of international standardized ratio (INR) and timely adjustment of warfarin dosage according to INR, which will result in difficult follow-up management, poor compliance, uncertainty of warfarin treatment effect, and even serious bleeding complications. According to relevant studies, the incidence of warfarin-related major bleeding is about 1%-2%, and the recurrence or aggravation of thrombus is also high. Rivaroxaban can simplify treatment, and is safe. It's also not easy to interact with food or drugs. Previous studies have shown that rivaroxaban is effective in preventing deep venous thrombosis after orthopaedic surgery. Rivaroxaban has also been shown to be safe and effective in anticoagulation therapy for patients with deep venous thrombosis and pulmonary embolism, and repeated coagulation monitoring is not required. However, Rivaroxaban lacks sufficient clinical data for perioperative adjuvant anticoagulation therapy of filter implantation. Therefore, this study should be carried out to provide the basis for DVT treatment guidelines and explore the clinical indications of rivaroxaban.

ELIGIBILITY:
Inclusion Criteria:

* Patients who was diagnosed with deep venous thrombosis of the lower extremity and implanted with a retrievable inferior vena cava filter.

Exclusion Criteria:

* Age < 18 years or age > 75 years,
* With obvious contraindications for anticoagulation therapy,
* Allergic to iodine contrast agents in the past,
* Pregnant or breastfeeding women,
* With malignant tumors and life expectancy < 1 year,
* Severe liver diseases (such as acute hepatitis, chronic active hepatitis or cirrhosis) or alanine aminotransferase levels were higher than three times the upper limit of normal.
* With other diseases that need anticoagulation,
* With previous heparin-induced thrombocytopenia,
* Bacterial endocarditis,
* Systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg,
* Taking cytochrome P450 3A4(CYP-450 3A4) inhibitors or inducers
* With severe renal insufficiency (creatinine clearance <30 mL/min)
* Allergic to the drug used in this study
* With permanent filter implantation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-05-08 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 4 months after the filter is retrieved
  Percentage of participants with all deaths
Pulmonary embolism related mortality | 4 months after the filter is retrieved
Percentage of Participants with bleeding | 4 months after the filter is retrieved
  Clinically relevant bleeding is defined as a composite of major or clinically relevant nonmajor bleeding
Percentage of Participants With Symptomatic Recurrent Venous Thromboembolism | 4 months after the filter is retrieved
  the Composite of Recurrent Deep Vein Thrombosis [DVT] or Fatal or Non-fatal Pulmonary Embolism [PE]

SECONDARY OUTCOMES:
Percentage of Participants With IVC Filter Retrieval Failure | 4 months after the filter is retrieved
  IVC filter retrieval failure is relevant to IVC filter complications (e.g. IVC thrombosis, IVC perforation, IVC filter migration or tilting and IVC filter embolization), system factors and technical factors.
Percentage of Participants With an Event for Net Clinical Benefit | 4 months after the filter is retrieved
  composite of primary efficacy outcomes and major bleeding, assessed in the intention-to-treat population.
Percentage of Participants With Other Vascular Events | 4 months after the filter is retrieved
  All pre-defined vascular events (ST segment elevation myocardial infarction, non ST segment elevation myocardial infarction, acute coronary syndrome, unstable angina, ischemic stroke, transient ischemic attack, pulmonary embolism, non-central nervous system systemic embolism or vascular death) will be assessed based results/films/images of confirmatory testing, and/or case summaries.

CONTACTS AND LOCATIONS:
Overall Officials: Zhejie Liu, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (7):
- China (7):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Yantai Yuhuangding Hospital, Yantai, Shangdong
  - Huadong Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanghai 5th People's Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - The second affiliated hospital of zhejiang university school of medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
Study protocol, statistical analysis plan and informed consent form will be openly available.

REFERENCES:
- [Background] Kearon C, Akl EA, Ornelas J, Blaivas A, Jimenez D, Bounameaux H, Huisman M, King CS, Morris TA, Sood N, Stevens SM, Vintch JRE, Wells P, Woller SC, Moores L. Antithrombotic Therapy for VTE Disease: CHEST Guideline and Expert Panel Report. Chest. 2016 Feb;149(2):315-352. doi: 10.1016/j.chest.2015.11.026. Epub 2016 Jan 7. PMID 26867832
- [Background] Jain A, Cifu AS. Antithrombotic Therapy for Venous Thromboembolic Disease. JAMA. 2017 May 16;317(19):2008-2009. doi: 10.1001/jama.2017.1928. No abstract available. PMID 28510665
- [Background] Breddin HK, Hach-Wunderle V, Nakov R, Kakkar VV; CORTES Investigators. Clivarin: Assessment of Regression of Thrombosis, Efficacy, and Safety. Effects of a low-molecular-weight heparin on thrombus regression and recurrent thromboembolism in patients with deep-vein thrombosis. N Engl J Med. 2001 Mar 1;344(9):626-31. doi: 10.1056/NEJM200103013440902. PMID 11228276
- [Background] Schulman S, Zondag M, Linkins L, Pasca S, Cheung YW, de Sancho M, Gallus A, Lecumberri R, Molnar S, Ageno W, Le Gal G, Falanga A, Hulegardh E, Ranta S, Kamphuisen P, Debourdeau P, Rigamonti V, Ortel TL, Lee A. Recurrent venous thromboembolism in anticoagulated patients with cancer: management and short-term prognosis. J Thromb Haemost. 2015 Jun;13(6):1010-8. doi: 10.1111/jth.12955. Epub 2015 May 9. PMID 25851122
- [Background] Turpie AG, Lassen MR, Davidson BL, Bauer KA, Gent M, Kwong LM, Cushner FD, Lotke PA, Berkowitz SD, Bandel TJ, Benson A, Misselwitz F, Fisher WD; RECORD4 Investigators. Rivaroxaban versus enoxaparin for thromboprophylaxis after total knee arthroplasty (RECORD4): a randomised trial. Lancet. 2009 May 16;373(9676):1673-80. doi: 10.1016/S0140-6736(09)60734-0. Epub 2009 May 4. PMID 19411100
- [Background] Lassen MR, Ageno W, Borris LC, Lieberman JR, Rosencher N, Bandel TJ, Misselwitz F, Turpie AG; RECORD3 Investigators. Rivaroxaban versus enoxaparin for thromboprophylaxis after total knee arthroplasty. N Engl J Med. 2008 Jun 26;358(26):2776-86. doi: 10.1056/NEJMoa076016. PMID 18579812
- [Background] Prins MH, Lensing AW, Brighton TA, Lyons RM, Rehm J, Trajanovic M, Davidson BL, Beyer-Westendorf J, Pap AF, Berkowitz SD, Cohen AT, Kovacs MJ, Wells PS, Prandoni P. Oral rivaroxaban versus enoxaparin with vitamin K antagonist for the treatment of symptomatic venous thromboembolism in patients with cancer (EINSTEIN-DVT and EINSTEIN-PE): a pooled subgroup analysis of two randomised controlled trials. Lancet Haematol. 2014 Oct;1(1):e37-46. doi: 10.1016/S2352-3026(14)70018-3. Epub 2014 Sep 28. PMID 27030066
- [Background] EINSTEIN Investigators; Bauersachs R, Berkowitz SD, Brenner B, Buller HR, Decousus H, Gallus AS, Lensing AW, Misselwitz F, Prins MH, Raskob GE, Segers A, Verhamme P, Wells P, Agnelli G, Bounameaux H, Cohen A, Davidson BL, Piovella F, Schellong S. Oral rivaroxaban for symptomatic venous thromboembolism. N Engl J Med. 2010 Dec 23;363(26):2499-510. doi: 10.1056/NEJMoa1007903. Epub 2010 Dec 3. PMID 21128814
- [Background] EINSTEIN-PE Investigators; Buller HR, Prins MH, Lensin AW, Decousus H, Jacobson BF, Minar E, Chlumsky J, Verhamme P, Wells P, Agnelli G, Cohen A, Berkowitz SD, Bounameaux H, Davidson BL, Misselwitz F, Gallus AS, Raskob GE, Schellong S, Segers A. Oral rivaroxaban for the treatment of symptomatic pulmonary embolism. N Engl J Med. 2012 Apr 5;366(14):1287-97. doi: 10.1056/NEJMoa1113572. Epub 2012 Mar 26. PMID 22449293
- [Derived] Zhang L, Li M, Zhu Y, Shi Z, Zhang W, Gao B, Li L, Fang Z, Yang G, Han W, Wang L, Yin L, Ke X, Yue J, Gu Z, Liu Z. Efficacy and safety of rivaroxaban in patients with inferior vena cava filter placement without anticoagulation contraindications (EPICT): a prospective randomised controlled trial study protocol. BMJ Open. 2021 Oct 25;11(10):e045530. doi: 10.1136/bmjopen-2020-045530. PMID 34697109